## GlaxoSmithKline Group of Companies

**Division:** World Wide Development **Retention Category:** GRS019

**Information Type:** Reporting and Analysis Plan

| Title: | Reporting and Analysis Plan for A Phase I Open-Label, Dose |
|--------|---------------------------------------------------------------|
| | Escalation Study to Investigate the Safety, Pharmacokinetics, |
| | Pharmacodynamics, and Clinical Activity of GSK2820151 in |
| | Subjects with Advanced or Recurrent Solid Tumors [Study |
| | 201893] |
| | • |

**Compound Number:** GSK2820151

**Effective Date:** 08-FEB-2019

Subject: Oncology, Reporting and Analysis Plan

## Author's Name, Title and Functional Area:

PPD

Principal Statistician, Biostatistics ICON Clinical Research

## Approved by:

PPD Date

Statistics Director Clinical Statistics (UK) RD Projects Clinical Platforms & Sciences GSK

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| ABE | BREVIA | TIONS | 4 |
|---|---|---|---|
| 1. | INTRO | DUCTION | 7 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4.<br>2.5. | ARY OF KEY PROTOCOL INFORMATION. Changes to the Protocol Defined Statistical Analysis Plan. Study Objective(s) and Endpoint(s). Statistical Hypotheses. Pharmacokinetic (PK) and PK/Pharmacodynamic Hypotheses. Study Design. | 8<br>9<br>9 |
| 3. | PLANN<br>3.1.<br>3.2. | NED ANALYSESInterim AnalysesFinal Analyses | .11 |
| 4. | SAMPI<br>4.1.<br>4.2. | LE SIZE CONSIDERATIONS | .12 |
| 5. | ANALY<br>5.1.<br>5.2.<br>5.3.<br>5.4. | /SIS POPULATIONS All Enrolled Population All Treated Population PK Population Analysis Datasets | .12<br>.12<br>.12 |
| 6. | TREAT<br>6.1. | TMENT COMPARISONS Data Display Treatment and Other Subgroup Descriptors | |
| 7. | GENE | RAL CONSIDERATIONS FOR DATA ANALYSES | .12 |
| 8. | DATA<br>8.1.<br>8.2. | HANDLING CONVENTIONS. Premature Withdrawal and Missing Data Derived and Transformed Data 8.2.1. Reference dates 8.2.2. Study Day for Safety Measures 8.2.3. Study Day for Efficacy 8.2.4. Duration and Elapsed Time 8.2.5. Imputation of Partial Dates 8.2.6. Imputation of Missing Exposure End Dates 8.2.7. Baseline Definition 8.2.8. Change from baseline 8.2.9. Multiple Assessments 8.2.10. Actual Treatment 8.2.11. Extended Loss to Follow-up or Extended Time without an Adequate Assessment 8.2.12. Date Associated with Response | .13<br>.13<br>.13<br>.13<br>.14<br>.14<br>.17<br>.17<br>.18<br>.18 |
| | 8.3. | Values of Potential Clinical Importance | .19 |

## 

| | | 8.3.2. | Vital Signs | 19 |
|---|---|---|---|---|
| 9. | STUD | Y POPUL | ATION ANALYSES | 20 |
| | 9.1. | Disposit | ion of Subjects | 20 |
| | 9.2. | | Deviations | |
| | 9.3. | | aphic and Baseline Characteristics | |
| | 9.4. | | ent Compliance | |
| | 9.5. | | itant Medications | |
| | 9.6. | | uent Anticancer Therapies | |
| 10. | EFFIC | CACY ANA | ALYSES | 21 |
| 11. | SAFE | TY ANAL | YSES | 23 |
| | 11.1. | | f Exposure | |
| | 11.2. | | Events | |
| | 11.3. | | Events of Special Interest | |
| | 11.4. | | and Serious Adverse Events (SAEs) | |
| | 11.5. | Adverse | Events Leading to Discontinuation of Study Treatment and/or | |
| | | Withdra | wal from the Study and Other Significant Adverse Events | 24 |
| | 11.6. | | Laboratory Evaluations | |
| | 11.7. | Other S | afety Measures | 25 |
| 12. | HEAL | TH OUT | COMES ANALYSES | 25 |
| 13. | PHAR | MACOKI | NETIC ANALYSES | 25 |
| | 13.1. | | ncentration Measures | |
| | 13.2. | | and Summarizing Pharmacokinetic Parameters | |
| 14. | PHAR | MACOGE | ENETIC DATA ANALYSES | 26 |
| 15. | REFE | RENCES | | 27 |
| 16. | APPE | NDIX 1: L | IST OF DATA DISPLAYS | 28 |
| | 16.1. | | splay Numbering | |
| | 16.2. | | ble | |
| | 16.3. | | ings | |
| | | | 4 Lietings | |

## **Abbreviations**

| 1,5 AG | 1,5 –Anhydroglucitol |
|---|---|
| ADaM | Analysis Data Model |
| AE(s) | Adverse event(s) |
| AESI | Adverse events of special interest |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| AUC | Area under the curve |
| AUC(0-∞) | Area under the curve from zero to infinity |
| AUC(0-τ) | Area under the plasma concentration-time curve |
| BET | Bromodomain & Extra-Terminal |
| BRD | Bromodomain |
| β-hCG | Beta-human chorionic gonadotropin |
| BUN | Blood urea nitrogen |
| Cav | Average observed concentration |
| CDISC | Clinical Data Interchange Standards Consortium |
| CK | Creatine kinase |
| CKMB | Creatine kinase MB isoenzyme |
| CL/F | Clearance |
| Cmax | Maximum observed concentration |
| CPMS | Clinical Pharmacology Modelling and Simulation |
| CR | Complete response |
| CRF | Case report form |
| CSR | Clinical Study Report |
| Ст | Trough concentration |
| CV | Cardiovascular |
| CV% | Percentage coefficient of variance |
| DLT | Dose-limiting toxicity |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| FTIH | First time in human |
| GSK | GlaxoSmithKline |
| HDL | High-density lipoprotein |
| HGB | Hemoglobin |
| ICH | International Council on Harmonization of Technical Requirements for |
| | Registration of Pharmaceuticals for Human Use |
| IDSL | Integrated Data Standards Library |
| IEC/IRB | Independent ethics committee/institutional review board |
| IL-6 | Interleukin 6 |
| INR | International normalized ratio |
| LDL | Low-density lipoprotein |
| LLN | Lower limit of normal |

## 

| LPS | Lipopolysaccharide |
|-----------|--------------------------------------------------------|
| LVEF | Left ventricular ejection fraction |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram(s) |
| msec | Millisecond(s) |
| MTD | Maximum tolerated dose |
| NCI-CTCAE | National Cancer Institute- Common Terminology Criteria |
| | for Adverse Events |
| N-CRM | Neuenschwander - Continuous Reassessment Method |
| NQ | Non-quantifiable |
| NT-proBNP | N-terminal pro–B-Type natriuretic peptide |
| ORR | Objective response rate |
| PD | Progressive disease |
| PFS | Progression free survival |
| PGx | Pharmacogenomics |
| PK | Pharmacokinetics |
| PR | Partial response |
| PT | Preferred term |
| PTT | Partial thromboplastin time |
| FACTS | Fixed and Adaptive Clinical Trial Simulator |
| QTc | Corrected QT interval |
| QTcF | Corrected QT (Fridericia's formula) |
| RAP | Reporting and Analysis Plan |
| RBC | Red Blood Cell |
| RECIST | Response criteria in solid tumors |
| Ro | The observed accumulation ratio |
| RP2D | Recommended Phase 2 dose |
| SAE(s) | Serious adverse event(s) |
| SOC | System organ class |
| SD | Stable disease |
| t½ | Apparent terminal phase half-life |
| tmax | Time to Cmax |
| TSH | Thyroid Stimulating Hormone |
| TTE | Time to event |
| ULN | Upper limit of normal |
| Vz/F | Volume of distribution |
| WBC | White blood cells |

201893

## **Trademark Information**

| Trademarks of the GlaxoSmithKline group of |
|--------------------------------------------|
| companies |
| NONE |

| Trademarks not owned by the GlaxoSmithKline group of companies |
|----------------------------------------------------------------|
| FACTS |
| SAS |

#### 1. INTRODUCTION

This reporting and analysis plan (RAP) details all planned analyses required for a Clinical Study Report of study 201893. This is a first time in human (FTIH), open-label, dose escalation study will assess the safety, pharmacokinetics (PK), pharmacodynamics, and preliminary clinical activity of GSK2820151 in subjects with advanced or recurrent solid tumors.

For further information on the study design, see Protocol Amendment dated 08-JUN-2017 (2014N215112\_04).

The RAP was written by staff of ICON Clinical Research. The execution of the RAP, with exception to Neuenschwander - Continual Reassessment Method (N-CRM) - based analyses using the Fixed and Adaptive Clinical Trial Simulator (FACTS), will be undertaken by staff of ICON Clinical Research.

All decisions regarding final analysis, as defined in this RAP document, have been made prior to Database Freeze of the study data. Effective November 17 2017, GSK has made the difficult decision to discontinue the development of GSK2820151 in solid tumors. This decision was made after careful consideration of the following factors:

- With the increasing amount of clinical data now available on Bromodomain & Extra-Terminal (BET) inhibitors, the opportunity for GSK2820151 to show a differentiated profile with significant additional clinical benefit has decreased.
- With more than 15 BET inhibitors in clinical development, it was very challenging to enroll to the BET inhibitor study (201893), which enrolled only 4 subjects over a period of 1.5 years.

At the time the study termination decision was made, one subject was still receiving treatment. The study terminated when the last subject completed last scan on November 18 2018 and showed disease progression. A total of 5 subjects have enrolled into the study.

Due to the early termination decision and the small number of subjects, only listings of the data will be generated.

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

| <b>Protocol Section</b> | Change from Protocol | Rationale |
|---|---|---|
| Section 11.4.2<br>Interim Analysis | No interim analysis in SAP | Sponsor made the decision to terminate the study early and no interim analysis needed |
| Section 11.2 Continual Reassessment Method | No N-CRM analysis in SAP | Sponsor made the decision to terminate the study early and did not get into N-CRM analysis phase |
| Section 11 Statistical Considerations and Data Analyses | No summary tables and figures No statistical analysis of pharmacokinetic parameters | Sponsor made the decision to terminate the study early and no tables/figures needed, only listings provided |
| Section 8.3.9 Clinical Safety Laboratory Assessments | No Creatinine Phosphokinase | This test was not collected per CRF |
| Section 11.5.3 Other Analyses | No biomarker,<br>pharmacodynamics exploratory<br>analyses performed | Sponsor made decision that biomarkers samples were not collected after 11Jan2018 and the biomarker samples collected by 11Jan2018 were destroyed. |

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary | |
| To determine the safety, tolerability and maximum tolerated dose (MTD) of GSK2820151 in subjects 18 years or older with advanced or recurrent solid tumors. | Adverse events (AEs), serious adverse events (SAEs), dose reductions or delays, withdrawals due to toxicities and changes in safety assessments (e.g., laboratory parameters, vital signs, electrocardiogram (ECG), cardiotoxicity, gastrointestinal, etc.) |
| Secondary | , <u>,</u> , |

| Objectives | Endpoints |
|---|---|
| To determine a recommended Phase 2 dose<br>(RP2D) of GSK2820151 in subjects 18 years or<br>older. | Safety profile (AEs, SAEs, dose-limiting toxicities [DLTs]), clinical response, and pharmacodynamics data |
| To characterize the PK of GSK2820151 in subjects 18 years or older. | PK parameter values for GSK2820151 following single and repeat-dose oral administration in subjects 18 years or older. |
| To evaluate the effect of treatment with GSK2820151 on tumor growth and subject survival. | Objective response rate (ORR) by various imaging modalities and progression free survival (PFS). |
| To evaluate cardiac safety, including the potential for corrected QT interval (QTc) prolongation, of GSK2820151 and to assess PK/QTc relationship. | Changes in cardiac safety including QTc following single and repeat-dose oral administration of GSK2820151. |
| Exploratory | |
| To evaluate the exposure response<br>(pharmacokinetic/pharmacodynamics [PK/PD])<br>relationship between GSK2820151 and safety<br>and efficacy parameters. | Dose-related change in molecular markers (e.g., gene transcription and/or expression of proteins regulated by BRD proteins) in peripheral blood samples. |
| To evaluate systemic and ex vivo on-target BET inhibitory effects | Changes from baseline and dose/response relationship in ex vivo lipopolysaccharide (LPS)-induced cytokines, including interleukin 6 (IL-6), in whole blood, and systemic cytokines, including IL-6. |
| To identify potential indicators of sensitivity or response to GSK2820151. | Transcriptomic studies of blood; correlation of baseline genetic and genomic profiles with response. |

## 2.3. Statistical Hypotheses

The primary endpoints of this study are safety and tolerability; the MTD and RP2D will also be determined. No formal statistical hypotheses will be tested. The primary focus will be on determining the recommended dose for further exploration, the safety profile, and the PK of GSK2820151 in subjects with advanced cancer. Analyses will be descriptive and exploratory.

## 2.4. Pharmacokinetic (PK) and PK/Pharmacodynamic Hypotheses

There is no formal statistical hypothesis for PK and pharmacodynamic analyses.

## 2.5. Study Design

This study is a single-agent, open-label, dose-escalation study to determine the MTD (and RP2D), based on the safety, pharmacokinetic, and pharmacodynamic profiles observed after oral administration of GSK2820151. Eligible subjects with advanced or recurrent solid tumors will be enrolled in the dosing cohorts until MTD is established. All subjects will receive study drug. Subjects may continue treatment in the study until disease progression, unacceptable toxicity, or withdrawal of consent (for specific stopping criteria, see Protocol Section 5.4). The duration of study will depend on recruitment rates and the timing of subjects' duration on study (withdrawal rates due to toxicity or progression).

This study will utilize an accelerated dose escalation phase in order to minimize suboptimal drug exposures, followed by a conventional 3+3 dose escalation phase to achieve MTD. Initially, one subject per dose cohort will be recruited (accelerated dose escalation phase) until the first instance of  $a \ge Grade\ 2$  drug related non-hematological

toxicity or dose-limiting toxicity (DLT, see Protocol Section 4.2.4). Further cohorts will be recruited in blocks of three subjects (3+3 dose escalation phase). Additional subjects may be enrolled at previously cleared dose levels in order to obtain further data for PK and/or pharmacodynamic analysis. Once MTD is determined, additional subjects (18 subjects total at MTD) may be enrolled to collect additional safety data (Figure 1). The total duration of study for each subject will be dependent upon the safety, tolerability and efficacy of GSK2820151.

In the accelerated dose escalation cohorts and the 3+3 dose escalation cohorts, the dose will be escalated based on PK data, the safety profile of the current and prior cohorts, as well as the predicted DLT rates on all potential doses from the N-CRM analysis [Neuenschwander, 2008]. N-CRM design is a type of Bayesian adaptive dose-escalation scheme (see Protocol Section 11.2). The method is fully adaptive and makes use of all the DLT information available at the time of each dose assignment. The DLT information of all subjects enrolled in the trial are used to update the estimated dose-toxicity relationship and provide supportive information in addition to the 3+3 design in the next escalation/de-escalation decision.

The RP2D will be determined based on the MTD or biologically active dose (example:clinical response), the safety profile, and available pharmacodynamic data generated from all subjects. If necessary alternate schedules can be explored to determine additional biologically active doses even after a RP2D is defined.



(Dose increase at any dose escalation will be ≤2 fold.)

Figure 1: Dose Escalation Scheme

Projected dose levels are 3 mg, 6 mg, 12 mg, 20 mg, 40 mg, 60 mg, 100 mg, 150 mg, 200 mg, and 300 mg. Additional doses and schedules may be explored based on emerging safety, PK, and pharmacodynamic data. Actual dose escalation doses and decisions, based on observed data, will be executed based on guidance described in Protocol Section 4.2.2 and Protocol Section 4.2.3.

The schedule for study assessments can be found in Protocol Section 8.

#### 3. PLANNED ANALYSES

In line with ICH E9 [European Agency for the Evaluation of Medicinal Products, 1998], membership of the analysis populations will be determined using the definitions in Section 5 of this RAP.

## 3.1. Interim Analyses

Interim PK data was reviewed at dose escalation meeting at each dose by GSK. Non Compartment analyses for Dose Escalation Cohorts was performed using Phoenix Winnonlin version 6.4 or higher under the supervision of clinical Pharmacology Modeling and Simulation (CPMS), GSK.

No N-CRM analysis was performed for the study due to the termination of the study.

## 3.2. Final Analyses

Final analyses will be performed after all subjects have permanently discontinued study treatment and the final study database is frozen.

See Sections 5 to 16 for details regarding the planned analyses and description of displays to be produced.

## 4. SAMPLE SIZE CONSIDERATIONS

## 4.1. Sample Size Assumptions

The total number of subjects to be enrolled into this study will depend on the number of subjects needed to characterize individual dose cohorts for the determination of the maximum tolerated dose of GSK2820151; the final sample size is not driven by statistical considerations. However, it is anticipated that approximately 30 to 50 subjects will be enrolled with a maximum of 80 subjects.

## 4.2. Sample Size Re-estimation or Adjustment

No sample size re-estimation will be performed.

#### 5. ANALYSIS POPULATIONS

## 5.1. All Enrolled Population

The **All Enrolled Population** is defined as all subjects who have consented to participate in the study and have not screen failed.

## 5.2. All Treated Population

The **All Treated Population** is defined as all subjects who receive at least one dose of GSK2820151. Safety and anti-cancer activity will be evaluated based on this analysis population.

## 5.3. PK Population

The **PK Population** will consist of all subjects from the All Treated Population for whom a PK sample is obtained and analysed.

## 5.4. Analysis Datasets

Analysis datasets will be created according to Clinical Data Interchange Standards Consortium (CDISC) version 3.1.3/ Analysis Data Model (ADaM) version 1.0 standards, and data will be listed according to GSK Integrated Data Standards Library (IDSL) reporting standards. Formatting for dates, times, and decimal places will follow GSK standards except where specified.

#### 6. TREATMENT COMPARISONS

There are no treatment comparisons in the study.

**6.1. Data Display Treatment and Other Subgroup Descriptors**Unless otherwise stated, all data will be pooled and listed by investigated GSK2820151 dose cohorts.

#### 7. GENERAL CONSIDERATIONS FOR DATA ANALYSES

SAS 9.3 or higher version will be used to perform all data analyses and generate listings. Data in the database will be presented in by-subject data listings.

#### 8. DATA HANDLING CONVENTIONS

## 8.1. Premature Withdrawal and Missing Data

Because study treatment is dependent on the study endpoints (e.g., progression, i.e. not a fixed treatment duration), the length of treatment for each subject will depend on the efficacy and toxicity of the treatment, so the duration of treatment will vary across subjects. Similarly the duration of follow up will also vary. All available PFS data will be analyzed using suitable statistical methods; subjects with shorter treatment and follow-up due to the natural history of their disease or medical necessities of the treatment of their disease will not be considered to have missing PFS data. For endpoints which determine the percentage of responders, subjects with unknown/not evaluable or missing best overall response will be assumed to be non-responders, and will be included in the denominator when calculating the percentages.

In the event that the study is terminated, all available data will be listed.

Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument. These data will be indicated by the use of a "blank" in subject listing displays. Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.

There will be no other imputation for missing data other than what's described in Section 8.2 for partial dates and for missing exposure end dates.

#### 8.2. Derived and Transformed Data

The following sections provide a general description of the derived and transformed variables used to describe and analyze the data. Separate analysis dataset specifications provide full details on all data derivations and transformations including descriptions of core standard algorithms and standard oncology algorithms. The analysis dataset specifications will clearly communicate the content and source of the datasets supporting the statistical analyses.

#### 8.2.1. Reference dates

Unless otherwise stated, the safety reference (start) date will be the start of treatment of GSK2820151. This will also be the efficacy reference date for this study. The reference date for baseline characteristics (e.g. age) will be the date of screening.

## 8.2.2. Study Day for Safety Measures

If the date of interest occurs on or after the safety reference date then the safety study day will be calculated as (date of interest - safety reference date) + 1. If the date of interest occurs before the safety reference date then the safety study day will be calculated as (date of interest-safety reference date). There is no safety study day 0.

## 8.2.3. Study Day for Efficacy

If the date of interest occurs on or after the efficacy reference date then efficacy study day will be calculated as (date of interest - efficacy reference date) + 1. If the date of interest occurs prior to the efficacy reference date

then efficacy study day will be calculated as (date of interest – efficacy reference date). There is no efficacy study day 0.

## 8.2.4. Duration and Elapsed Time

Durations (e.g., the duration of an AE, duration of exposure, etc.) are calculated as the stop date minus the start date plus one.

For elapsed time (e.g., the time since initial diagnosis):

- If the reference date is on or after the event date, then the elapsed time is the reference date minus the event date + 1.
- If the reference date is before the event date then the elapsed time is the reference date minus the event date.

When reporting time to event (TTE) durations in months, divide the number of days by 30.4375; to report in weeks divide the number of days by 7; to report in years divide the number of days by 365.25. These algorithms for time to event return decimal numbers, and ignore the actual numbers of days in the months or years between start date and stop date. The "year" used in these algorithms is 365.25 days long, and the "month" is one twelfth of that year.

## 8.2.5. Imputation of Partial Dates

Imputed partial dates will not be used to derive study day, duration (e.g., duration of AEs), or elapsed time variables. In addition, imputed dates are not used for deriving the last contact date in progression free survival analysis dataset.

Imputed dates will not be displayed in listings. However, where necessary, display macros may impute dates as temporary variables for the purpose of sorting data in listings only. Partial dates may be imputed as outlined below.

The partial date imputation will follow ADaM conventions. The ADaM approach is to populate the numeric date variables with the imputed date and add a flag variable to the dataset that indicates the level of imputation.

The flag variable can contain the values: blank, 'D', 'M', 'Y'.

blank: indicates that no imputation was done

D='Day': indicates that the day portion of the date is imputed

M='Month': indicates that the month and day portions of the date are imputed

Y='Year': indicates that the entire date (year, month, and day) is imputed

Example of Date Variables:

XYZD - character date variable

XYZDT - numeric date variable

XYZDTFL - flag variable

Details on imputing partial dates for specific datasets are outlined below.

## **Adverse Events (AE):**

Imputations in the adverse events dataset are used for slotting events to the appropriate study time periods and for sorting in data listings.

| Dataset | Date | Missing<br>Element | Rule |
|---|---|---|---|
| Adverse<br>Events<br>(AE) | Start<br>Date | day,<br>month,<br>and year | No Imputation for completely missing dates |
| | | day,<br>month | <ul> <li>If study treatment start date is missing (i.e. subject did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> <li>If study treatment start date is missing (i.e. subject did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = 1st of month.</li> </ul> </li> </ul> |
| | | | <ul> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> |
| | End<br>Date | | No imputation for partial end dates will be performed |

# Anticancer Therapy and Radiotherapy, Surgery, Concomitant Medication and Blood and Blood Supportive Care Products:

Start dates are generally not imputed. If start dates need to be imputed for sorting in data listings, the rules of imputation is defined as below:

| Dataset | Date | Missing<br>Element | Rule |
|---|---|---|---|
| Anticancer<br>Therapy | Start<br>Date | day,<br>month, and<br>year | No Imputation for completely missing dates |
| Radiotherapy | | day, month | • If partial date contains a year only set to January 1st. |
| Surgical<br>Procedures | | day | If partial date contains a month and year set to the 1st of the month. |
| Concomitant<br>Medication | | | |
| Blood and Blood<br>Supportive Care<br>Products | | | |

#### **Time to Event and Overall Response:**

Start dates for follow-up anticancer therapy, radiotherapy (where applicable), and surgical procedures (where applicable) will be temporarily imputed in order to define event and censoring rules for progression-free survival, response rate, or duration of response (i.e. start date for new anticancer therapy). Dates will only be imputed when a month and year are available but the day is missing. The imputed date(s) will not be stored on the anticancer therapy, radiotherapy, or surgical procedure datasets. The following rules will be used to impute the date when partial start dates are present on anticancer therapy radiotherapy, and/or surgical procedures dataset[s]:

| Dataset | Date | Missing<br>Element | Rule |
|---|---|---|---|
| Anticancer<br>Therapy | Start<br>Date | day, month, and year | No Imputation for completely missing dates |
| Where applicable: | | | |
| Radiotherapy | | | |
| Surgical<br>Procedures | | | |

| Dataset | Date | Missing<br>Element | Rule |
|---|---|---|---|
| | | day, month | No imputation for missing day and month (note the eCRF should only allow for missing day) |
| | | day | <ul> <li>If partial date falls in the same month as the last dose of study treatment, then assign to earlier of (date of last dose of study treatment+1, last day of month).</li> <li>If partial date falls in the same month as the subject's last assessment and the subject's last assessment is PD, then assign to earlier of (date of PD+1, last day of month).</li> <li>If both rules above apply, then assign to latest of the 2 dates</li> <li>Otherwise, impute missing day to the first of the month.</li> </ul> |
| | End<br>Date | | No imputation for partial end dates will be performed |

The date of new anticancer therapy is derived as the earliest date of new anticancer therapy (e.g., chemotherapy), radiotherapy (where applicable), or cancer related surgical procedure (where applicable) and will include imputed dates.

## 8.2.6. Imputation of Missing Exposure End Dates

In general, completely missing dates are not imputed. However, subjects in oncology trials may still be on study treatment when analyses are performed and so may have missing exposure end dates in their last dosing record. Missing exposure end dates will be imputed. For subjects with missing exposure end dates at the time of data cutoff, the exposure end date will be imputed to the earliest of: the date of the data cutoff, the date of withdrawal from the study, or the death date. The imputed exposure end date will be used to calculate cumulative dose and exposure duration. Imputed exposure end dates will be stored on the study treatment end date variable.

#### 8.2.7. Baseline Definition

Baseline will be defined as the most recent, non-missing value prior to or on the first study treatment dose date for GSK2820151. For laboratory data, baseline will be defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. If there are no central labs collected for a subject and lab test prior to or on the first dose of study treatment, the most recent, non-missing value from a local laboratory prior to or on the first dose of study treatment will be defined as the baseline value.

If the latest pre-dose value is collected on the day of treatment, the time of treatment will be used to identify the baseline value. If the pre-dose time point value is identified as baseline, and the data is recorded in triplicate the average will be used.

For subjects who did not receive study treatment during the study, baseline will be defined as the latest, non-missing collected value.

## 8.2.8. Change from baseline

Change from baseline will be presented for ECG and ECOG data as described in Section 11.

Change from baseline is calculated as:

• For records occurring after baseline: (visit value) – baseline value.

For the triplicate measurements, the average value will be used as visit value.

Unless otherwise stated, if either the baseline or visit value is missing, the change from baseline and/or percent change from baseline is set to missing as well.

## 8.2.9. Multiple Assessments

Data from all assessments (scheduled and unscheduled), including multiple assessments, will be included in listings.

#### 8.2.10. Actual Treatment

A subjects' actual treatment will be derived from exposure data.

#### 8.2.11. Extended Loss to Follow-up or Extended Time without an Adequate Assessment

If two or more scheduled disease assessments are missed and are then followed by an assessment of progressive disease (PD) or death, PFS will be censored at the last adequate assessment prior to PD or death. As the scheduled disease assessment is every 8 weeks, a window of 119 days (16 weeks + 7 day window) will be used to determine whether there was an extended time without adequate assessment. That is, if the time difference between PD/death and last adequate assessment is more than 119 days, then PFS will be censored at the last adequate assessment prior to PD/death.

#### 8.2.12. Date Associated with Response

For each disease assessment after baseline, a date will be associated with the response based on collective group of disease assessments made within the protocol visit window. For complete response (CR) and partial response (PR), this will be assigned to the latest date within the disease assessments. For stable disease (SD), Non-CR/Non-PD or Not Evaluable, this will be assigned to the earliest date within the disease assessments. For PD, assign to the earliest assessment date associated with the progression.

## 8.3. Values of Potential Clinical Importance

## 8.3.1. Laboratory Parameters

Reference ranges for all laboratory parameters collected throughout the study are provided by the laboratory. A laboratory value that is outside the reference range is considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Note: a high abnormal or low abnormal laboratory value is not necessarily of clinical concern. The laboratory reference ranges will be provided on the listings of laboratory data. Clinical laboratory test results outside of the reference range will be flagged in the listings.

To identify laboratory values of potential clinical importance, National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03 [NCI-CTCAE, 2010]) will be used to assign grades to the relevant laboratory parameters.

## 8.3.2. Vital Signs

To identify heart rate values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with the grades for 'Sinus bradycardia', 'Sinus tachycardia', 'Supraventricular tachycardia', and 'Ventricular tachycardia'.

The following criteria will be used to flag vital sign values that are values of potential clinical importance:

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|---|---|---|
| Decrease from baseline Heart Rate | Decrease to <60 | bpm |
| Increase from baseline Heart Rate | Increase to >100 | bpm |

To identify blood pressure values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with the grades for 'Hypertension'.

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|--------------------------|-------------------------------------------|------|
| Increase from baseline | ≥120 to <140 (Grade 1) | mmHg |
| Systolic Blood Pressure | ≥140 to <160 (Grade 2) | |
| | ≥160 (Grade 3) | |
| Increase from baseline | ≥80 to <90 (Grade 1) | mmHg |
| Diastolic Blood Pressure | ≥90 to <100 (Grade 2) | |
| | ≥100 (Grade 3) | |

Systolic blood pressure below 120 mmHg and diastolic blood pressure below 80 mmHg are considered as normal range and will receive Grade 0 designations.

To identify temperature values of potential clinical importance, NCI-CTCAE v4.03 will be used to assign categories that align with the grades for 'Hypothermia' and 'Fever'.

| Vital Sign Parameter | Potential Clinical Importance (PCI) Range | Unit |
|---|---|---|
| Increase from baseline temperature | Increase to ≥38 | Degrees C |
| Decrease from baseline temperature | Decrease to ≤35 | Degrees C |

#### 9. STUDY POPULATION ANALYSES

Unless otherwise stated, all data listings in this section will be based on the All Treated Population.

## 9.1. Disposition of Subjects

A listing of reasons for study withdrawal will be generated. A listing of study treatment discontinuation will be generated. The listing will include last dose date, and reasons for study treatment discontinuation.

#### 9.2. Protocol Deviations

All protocol deviations will be listed. A separated listing of inclusion/exclusion deviations will also be provided.

## 9.3. Demographic and Baseline Characteristics

The demographic characteristics (e.g., age, sex, ethnicity, race, baseline height, and baseline weight, body mass index) will be listed.

Race and racial combinations, and family history will be listed.

Disease characteristics, as well as these medical conditions, will be presented in data listings.

Prior anti-cancer therapy will be coded using GSK Drug coding dictionary and listed. A listing of prior anti-cancer therapy will show the relationship between Anatomical Therapeutic Chemical (ATC) Level 1, Ingredient, and verbatim text.

Prior anti-cancer radiotherapy will be listed. Prior cancer and non-cancer related surgeries will be listed.

## 9.4. Treatment Compliance

A listing of scheduled and actual treatments will be produced.

#### 9.5. Concomitant Medications

Concomitant medications will be coded using GSK Drug coding dictionary and listed. Listing for blood products or blood supportive care products will be provided.

## 9.6. Subsequent Anticancer Therapies

Follow-up anticancer therapy will be coded using GSK Drug coding dictionary. A data listing for follow up anticancer therapy will be provided.

Any follow-up anticancer surgeries will be listed.

#### 10. EFFICACY ANALYSES

The evaluation of anticancer activity will be evaluated based on the All Treated Population as defined in Section 5 unless otherwise specified. Since this is a Phase I study, anticancer activity will be evaluated based on clinical evidence and response criteria. Due to the very limited number of subjects, ORR was not calculated. It can be counted from the investigator assessed response listings if need.

## **Lesion Assessment and Response**

Lesion assessment method and timing, evaluation of disease, disease progression and response criteria will be conducted according to Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) [Eisenhauer EA. etc, 2009] as outlined in Appendix 8 of the protocol. Data listings for response will be provided.

## **Progression-Free Survival (PFS)**

PFS is defined as the interval of time (in weeks) between the start date of treatment and the earlier of the date of disease progression and the date of death due to any cause. Disease progression will be based on the assessments by the Investigator.

The date of documented disease progression will be defined as the date of disease progression based on eCRF entries. If an assessment occurs over multiple days, the earliest date of progression will be used. The date of death should be taken from the Record of Death page. Death on study due to any cause will be included.

If there is no adequate baseline assessment, the subjects will be censored at their start date of treatment. Subjects without any adequate post-baseline tumor assessments will be censored at the start date of treatment. If the subject received subsequent anti-cancer therapy prior to the date of documented events, PFS will be censored at the last adequate assessment (e.g. assessment where visit level response is CR, PR, or SD) prior to the initiation of therapy. Progressive disease (PD) will also be defined per RECIST 1.1 criteria. Otherwise, if the subject does not have a documented date of events, PFS will be censored at the date of the last adequate assessment.

Subjects who progressed or died after an extended period without adequate assessment will be censored at their date of last adequate assessment prior to progression or death even if subsequent information is available regarding progression or death. The date of response at that assessment will be used for censoring. As the assessment schedule may change through the course of the protocol, specific rules for identifying extended loss to follow-up or extended time without an adequate assessment are provided in Section 8.2.11.

For subjects who receive subsequent anticancer therapy the following rules will apply:

• If the start date of the anticancer therapy is partial (i.e. either missing the day but has the month and year available or missing both day and month), the imputation rules described in Section 8.2.5 will be applied. No imputation will be made for completely missing dates.

• If anticancer therapy is started without documented disease progression or is started prior to documented disease progression, then PFS will be censored at the date of the last adequate assessment that is no later than the date of initiation of anticancer therapy (i.e. if an assessment occurs on the same day as the start of new anticancer therapy the assessment will be used - as it will be assumed the assessment occurred prior to the administration of new anticancer therapy). The date of response at the last adequate assessment will be used as the censoring value.

A summary of the assignments for progression and censoring dates for PFS are specified in the following table.

Table 1. Assignments for Progression and Censoring Dates for PFS Analysis

| Situation | Date of Event<br>(Progression/Death) or<br>Censoring | Outcome<br>Event (Progression/Death)<br>Or Censored |
|---|---|---|
| No (or inadequate) baseline tumor assessments and the subject has not died (if the subject has died follow the rules for death indicted at the bottom of the table) | Start Date of Treatment | Censored |
| No post-baseline assessments and the subject has not died (if the subject has died follow the rules for death indicted at the bottom of the table) | Start Date of Treatment | Censored |
| Progression documented between scheduled visits | Date of assessment of progression <sup>1</sup> | Event |
| No progression (or death) and no initiation of new anti-cancer therapy | Date of last 'adequate' assessment of response <sup>2</sup> | Censored |
| Received subsequent anti-cancer therapy prior to the date of documented events | Date of last 'adequate' assessment of respnose <sup>2,3</sup> (prior to starting initiation of therapy) | Censored |
| Received subsequent anti-cancer therapy prior to any adequate assessment | Start Date of Treatment | Censored |
| Received subsequent anti-cancer therapy and no progression (or death) | Date of last 'adequate' assessment of respnose <sup>2,3</sup> (prior to starting initiation of therapy) | Censored |
| Death or progression after more than one missed visit | Date of last 'adequate' assessment of response <sup>2</sup> (prior to missed assessments) | Censored |
| Death | Date of Death | Event |

- 1. The earliest of (i) Date of radiological assessment showing new lesion (if progression is based on new lesion); or (ii) Date of radiological assessment showing unequivocal progression in non-target lesions, or (iii) Date of last radiological assessment of measured lesions (if progression is based on increase in sum of measured lesions)
- 2. An adequate assessment is defined as an assessment where the Investigator determined response is CR, PR, or SD.
- 3. If PD and New anti-cancer therapy occur on the same day assume the progression was documented first e.g., outcome is progression and the date is the date of the assessment of progression). If anti-cancer therapy is started prior to any adequate assessments, censoring date should be the start date of treatment.

#### 11. SAFETY ANALYSES

Unless otherwise specified, all the safety analyses will be based on the All Treated Population as defined in Section 5.

#### 11.1. Extent of Exposure

Extent of exposure to GSK2820151 will be listed. The subject's average daily dose, defined as the cumulative dose divided by the duration of exposure for each subject, will be listed.

All dose reductions and dose interruptions will be listed separately.

#### 11.2. Adverse Events

AEs will be coded to the preferred term (PT) level using the Medical Dictionary for Regulatory Affairs (MedDRA dictionary version 21.1) and grouped by system organ class (SOC). AEs will be graded by the investigator according to the NCI-CTCAE v4.03.

All AEs will be listed.

## 11.3. Adverse Events of Special Interest

For any cardiovascular events detailed in Protocol Appendix 6 and all deaths, whether or not they are considered SAEs, specific Cardiovascular (CV) and Death sections of the eCRF will be required to be completed. These sections include questions regarding cardiovascular (including sudden cardiac death) and non-cardiovascular death. CV and death data will be listed separately.

## 11.4. Deaths and Serious Adverse Events (SAEs)

In the event that a subject has withdrawn consent, no data after the withdrawal of consent date from this subject including death is supposed to appear in the database, which should be part of the data cleaning process. A listing will be generated to provide subject-specific details on subjects who died.

SAEs are included in the listing of all adverse events. Separate supportive listings with subject-level details will be generated for

- Fatal SAEs
- Non-Fatal SAEs.

Primary and secondary cause of death will be presented in subject data listings.

# 11.5. Adverse Events Leading to Discontinuation of Study Treatment and/or Withdrawal from the Study and Other Significant Adverse Events

Separate AEs supportive listings will be generated with subject level details for those subjects:

- AEs leading to discontinuation of study treatment
- AEs leading to withdrawal from the study
- AEs leading to dose interruptions
- AEs leadings to dose reductions

## 11.6. Clinical Laboratory Evaluations

The assessment of laboratory toxicities will examine the following laboratory tests:

Clinical Chemistry: Total and direct bilirubin, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase, Total Protein, Albumin, Sodium, Potassium, Calcium, Blood Urea Nitrogen (BUN), Creatinine, Chloride, Fasting Glucose, Ionized Calcium, Gamma-glutamyltransferase, Total carbon dioxide, Uric Acid, and Magnesium.

**Hematology**: Hemoglobin (HGB), Platelet count, Red Blood Cell (RBC) count, White Blood Cell (WBC) count, Neutrophils (Absolute), Lymphocytes (Absolute), Monocytes (Absolute), Eosinophils (Absolute), Basophils (Absolute), Neutrophils (%), Lymphocytes (%), Monocytes (%), Eosinophils (%) and Basophils (%).

Thyroid Function Test: Thyroid-stimulating hormone (TSH) and free thyroxine (T4 and T3) test.

Urinalysis: pH, Microscopic examination, Specific gravity, Ketones, Protein, Glucose, Blood.

**Coagulation Test**: Prothrombin Time, Partial Thromboplastin Time (PTT), International Normalized Ratio (INR), and Fibrinogen.

**Pancreatic Markers**: Amylase, Lipase.

**Lipid Panel**: Triglycerides, Total Cholesterol, low density lipoprotein (LDL), and high density lipoprotein (HDL).

**Serum**: Creatine Kinase (CK), Creatine Kinase-MB isoenzyme (CKMB), Troponin I, Troponin T, N-terminal pro–B-Type natriuretic peptide (NT-proBNP), Thyroid-stimulating hormone (TSH), C-Peptide, 1,5-Anhydroglucitol (1,5 AG), Hemoglobin A1C, and Insulin.

Laboratory grades will be reported, where applicable, using the Common Terminology Criteria for Adverse Events (CTCAE v4.03). Listings of laboratory data will be provided.

## 11.7. Other Safety Measures

#### **Vital Signs**

A listing will be provided. Categories defined in Section 8.3.2 will be presented in the listing as well.

#### **Performance Status**

ECOG performance status will be listed. Change from baseline will be presented in the listing as well.

#### **ECG**

Listings of abnormal ECG findings and a listing of ECG values will be provided.

#### Left ventricular ejection fraction (LVEF)

LVEF results will be listed with subject level details including absolute change from baseline.

#### 12. HEALTH OUTCOMES ANALYSES

No health outcomes analyses were planned for the study.

## 13. PHARMACOKINETIC ANALYSES

PK analysis of GSK2820151 drug concentration-time data and derivation of PK parameters will be conducted by non-compartmental methods using Phoenix WinNonlin Version 6.4 or higher under the direction of Clinical Pharmacology Modelling and Simulation (CPMS), GSK. Unless otherwise stated, all listings in this section will be based on the Pharmacokinetic population.

## 13.1. Drug Concentration Measures

Drug concentration-time data will be listed for each subject.

## 13.2. Deriving and Summarizing Pharmacokinetic Parameters

For subjects in the active treatment group, the pharmacokinetic parameters will be determined directly from the concentration-time data and will be extracted from the pharmacokinetic concentration file by CPMS GSK.

For the calculation of individual pharmacokinetic profiles, if one or more non-quantifiable (NQ) values occur in a profile before the first measurable concentration, they will be assigned a value of zero concentration. If a single NQ value occurs between measurable concentrations in a profile, the NQ should generally be omitted (set to missing) in the derivation of pharmacokinetic parameters. If two or more NQ values occur in succession between measurable concentrations, these NQs and any subsequent measurable concentrations will be omitted (set to missing) for the derivation of pharmacokinetic parameters.

NQs which occur after the last measurable concentration will be omitted (set to missing) in the derivation of pharmacokinetic parameters.

The following PK parameters will be determined if data permit:

- maximum observed concentration (Cmax)
- time to Cmax (tmax)
- area under the plasma concentration-time curve (AUC(0-t), AUC(0- $\infty$ ) (Week1 Day1 only), AUC(0- $\tau$ ))
- apparent terminal phase half-life  $(t^{1/2})$
- Trough concentration ( $C\tau$ )
- The observed accumulation ratio (Ro)
  - The ratio of AUC(0- $\tau$ ) on Week 3 Day 4 / Week 1 Day 1 AUC(0- $\tau$ ) will be calculated to assess time invariance.
- Clearance (CL/F) and Volume of distribution (Vz/F)

All derived PK parameters will be listed.

## 14. PHARMACOGENETIC DATA ANALYSES

Further details on PGx analyses discussed in the protocol may be identified/addressed in a separate RAP, if applicable.

## 15. REFERENCES

Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, et al. New response evaluation criteria in solid tumors: Revised RECIST guidelines (version 1.1). Eur J Cancer. 2009; 45: 228-247.

NCI-CTCAE (NCI Common Terminology Criteria for Adverse Events), Version 4.03, DCTD, NCI, NIH, DHHS, June 14, 2010.

Neuenschwander B, Branson M, Gsponer T. Critical aspects of the Bayesian approach to phase I cancer trials. *Statistics Med.* 2008; 27:2420-2439.

## 16. APPENDIX 1: LIST OF DATA DISPLAYS

## 16.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Listings |
|------------------|----------|
| ICH Listings | 1 to 46 |
| Non-ICH Listings | 47 to 53 |

## 16.2. Deliverable

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

## 16.3. ICH Listings

| No. | Population | Title | Programming Notes | Deliverable |
|---|---|---|---|---|
| Subje | Subject Disposition | | | |
| 1. | All Treated | Listing of Subject Consent | ICH E3 | SAC |
| 2. | All Treated | Listing of Scheduled and Actual Treatment | ICH E3 | SAC |
| 3. | All Treated | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 4. | All Treated | Listing of GSK2820151 Treatment Discontinuations | ICH E3 | SAC |
| Proto | col Deviations | | | |
| 5. | All Treated | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| 6. | All Treated | Listing of Protocol Deviations | | |
| Demo | ographic and Ba | seline Characteristics | | |
| 7. | All Treated | Listing of Demographic Characteristics | ICH E3 | SAC |
| 8. | All Treated | Listing of Race | ICH E3 | SAC |
| 9. | All Treated | Listing of Family History | ICH E3 | SAC |
| 10. | All Treated | Listing of Medical Conditions | ICH E3 | SAC |
| 11. | All Treated | Listing of Disease Characteristics at Initial Diagnosis | ICH E3 | SAC |
| 12. | All Treated | Listing of Disease Characteristics at Screening | ICH E3 | SAC |
| Prior | Prior and Concomitant Medications | | | |
| 13. | All Treated | Listing of Prior Anti-Cancer Therapy | Study specific | SAC |
| 14. | All Treated | Listing of Prior Anti-Cancer Radiotherapy | Study specific | SAC |

| No. | Population | Title | Programming Notes | Deliverable |
|---|---|---|---|---|
| 15. | All Treated | Listing of Prior Cancer and Non-Cancer Related Surgical Procedures | Study specific | SAC |
| 16. | All Treated | Listing of Concomitant Medications | ICH E3 | SAC |
| 17. | All Treated | Listing of Blood Products and Blood Supportive Care Products | Study specific | SAC |
| 18. | All Treated | Listing of Follow-Up Anti-Cancer Therapy | Study specific | SAC |
| 19. | All Treated | Listing of Follow-Up Surgical Procedures | Study specific | SAC |
| Expo | sure and Treatn | nent Compliance | | |
| 20. | All Treated | Listing of Exposure to GSK2820151 | ICH E3 | SAC |
| 21. | All Treated | Listing of Dose Interruptions | ICH E3 | SAC |
| 22. | All Treated | Listing of Dose Reductions | ICH E3 | SAC |
| Adve | rse Events | | | |
| 23. | All Treated | Listing of Adverse Events Profiles | ICH E3 | SAC |
| Serio | us and Other Si | gnificant Adverse Events | | |
| 24. | All Treated | Listing of Fatal Serious Adverse Events | ICH E3 | SAC |
| 25. | All Treated | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC |
| 26. | All Treated | Listing of Adverse Events Leading to Discontinuations of GSK2820151 Treatment Profiles | ICH E3 | SAC |
| 27. | All Treated | Listing of Adverse Events Leading to Dose Interruptions | ICH E3 | SAC |
| 28. | All Treated | Listing of Adverse Events Leading to Dose Reductions | ICH E3 | SAC |
| 29. | All Treated | Listing of Adverse Events Recorded as Dose-<br>Limiting Toxicities | Study specific | SAC |
| 30. | All Treated | Listing of Adverse Events of Special Interest | Study specific | SAC |
| 31. | All Treated | Listing of Deaths | ICH E3 | SAC |
| 32. | All Treated | Listing of Subject Numbers for Specific Causes of Deaths | ICH E3 | SAC |
| All La | aboratory | | | |
| 33. | All Treated | Listing of Clinical Chemistry Data | ICH E3 | SAC |
| 34. | All Treated | Listing of Hematology Data | ICH E3 | SAC |
| 35. | All Treated | Listing of Thyroid Function Test Data | ICH E3 | SAC |
| 36. | All Treated | Listing of Urinalysis Data | ICH E3 | SAC |
| 37. | All Treated | Listing of Coagulation Data | ICH E3 | SAC |

| No. | Population | Title | Programming Notes | Deliverable |
|---|---|---|---|---|
| 38. | All Treated | Listing of Pancreatic Markers Data | ICH E3 | SAC |
| 39. | All Treated | Listing of Lipid Panel Data | ICH E3 | SAC |
| 40. | All Treated | Listing of Serum Data | ICH E3 | SAC |
| Vital | Signs | | | |
| 41. | All Treated | Listing of Vital Signs | ICH E3 | SAC |
| ECO | ECOG | | | |
| 42. | All Treated | Listing of ECOG Performance Status Scale | ICH E3 | SAC |
| ECG | ECG and LVEF | | | |
| 43. | All Treated | Listing of Abnormal ECG Findings | ICH E3 | SAC |
| 44. | All Treated | Listing of ECG Values | ICH E3 | SAC |
| 45. | All Treated | Listing of Change from Baseline ECG Values | ICH E3 | SAC |
| 46. | All Treated | Listing of Left Ventricular Ejection Fraction (LVEF) ECHO Results | ICH E3 | SAC |

## 16.4. Non-ICH Listings

| No. | Population | Title | Programming Notes | Deliverable |
|---|---|---|---|---|
| Effica | Efficacy Endpoints | | | |
| 47. | All Treated | Listing of Investigator-Assessed Response (RECIST 1.1) | Study specific | SAC |
| 48. | All Treated | Listing of Investigator–Assessed Target Lesions (RECIST 1.1) | Study specific | SAC |
| 49. | All Treated | Listing of Investigator–Assessed Non-Target Lesions (RECIST 1.1) | Study specific | SAC |
| 50. | All Treated | Listing of Investigator–Assessed New Lesions | Study specific | SAC |
| 51. | All Treated | Listing of Progression Free Survival (RECIST 1.1) | Study specific | |

## 

| No. | Population | Title | Programming Notes | Deliverable |
|---|---|---|---|---|
| Phari | Pharmacokinetic | | | |
| 52. | PK Population | Listing of GSK2820151 Pharmacokinetic Concentration-Time Data | ICH E3 | SAC |
| 53. | PK Population | Listing of Derived GSK2820151 Pharmacokinetic Parameters | ICH E3 | SAC |

## 201893

Protocol: GSK201893 Population: All Treated Page X of Y

Listing 1
Listing of Subject Consent

Country: xxxxxx

Investigator: xxxxx xxxxxx

| | Original Informed Consent | | | | Reconsented | | Pharmacogenetic Research Consent | | |
|---|---|---|---|---|---|---|---|---|---|
| Center/<br>Subject ID | Date | Consent<br>Version | Protocol<br>Version | Date | Consent<br>Version | Protocol<br>Version | Date | Reason | Date of<br>Withdrawal |
| xxxx/<br>xxxxxx | ddMMMyyyy | XXX | XXX | ddMMMyyyy | XXX | XXX | ddMMMyyyy | | |
| xxxx/<br>xxxxxx | ddMMMyyyy | xxx | XXX | ddMMMyyyy | XXX | xxx | | xxx | |
| xxxx/<br>xxxxxx | ddMMMyyyy | XXX | XXX | ddMMMyyyy | XXX | XXX | ddMMMyyyy | | ddMMMyyyy |

## 201893

Protocol: GSK201893
Population: All Treated
Page X of Y

#### Listing 2 Listing of Scheduled and Actual Treatment

Country: xxxxxx Center: XXXX

Investigator: xxxxxx xxxxxx

| Subject ID | Planned Treatment | Actual Treatment |
|------------|-------------------|------------------|
| | 2 | 2 |
| XXXX | 3 mg | 3 mg |
| | 6 mg | 6 mg |

## 201893

Protocol: GSK201893
Population: All Treated
Page X of Y

# Listing 3 Listing of Reasons for Study Withdrawal

| Treatment = GSK28201 | 3 | _ | | |
|---|---|---|---|---|
| Center/ | Date of | Study | | |
| Subject ID | Withdrawal | Day | Primary Reason | Subreason |
| xxxx/ | ddMMMyyyy | X | Study closed/terminated | I |
| xxxxxx | 222 | | <b>.</b> | |
| xxxx/ | ddMMMyyyy | X | Lost to Follow-up | |
| XXXXXX | | | | |
| xxxx/ | ddMMMyyyy | XX | Investigator discretion | |
| XXXXXX | | | | |

## 201893

Protocol: GSK201893
Population: All Treated

## Listing 4 Listing of GSK2820151 Treatment Discontinuations

| Center/ | Cumulative | Date of | Study | Primary Reason for |
|---|---|---|---|---|
| Subject ID | Dose (mg) | Last Dose | Day | Treatment Discontinuation |
| xxxxx/ | XXX | ddMMMyyyy | XX | xxxxxxxxxxxxx |
| XXXXXX | | 1 12500 | | |
| xxxxx/<br>xxxxxx | XXX | ddMMMyyyy | XX | XXXXXXXXXXXXXX |
| xxxxx/ | xxx | ddMMMyyyy | XX | xxxxxxxxxxxxx |
| XXXXXX | | | | |
| xxxxx/ | XXX | ddMMMyyyy | XX | Xxxxxxxxxxxxx |
| XXXXXX | | | | |

## 201893

Protocol: GSK201893
Population: All Treated

| Listing | 5 |
|---------|---|
|---------|---|

Listing of Subjects with Inclusion/Exclusion Criteria Deviations

Treatment = xxxxxx

| Center/<br>Subject ID | Туре | Criterion |
|---|---|---|
| xxxxx/<br>xxxxxx | Inclusion | Written informed consent provided |
| xxxxx/<br>xxxxxx | Exclusion | Prior malignancy of the central nervous system or malignancies related to human immunodeficiency virus (HIV) or solid organ transplant |
| xxxxx/<br>xxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
# 201893

Protocol: GSK201893
Population: All Treated

# Listing 6 Listing of Protocol Deviations

| Treatment = xxx | <pre>Ireatment = xxxxxx</pre> | | |
|---|---|---|---|
| Center/<br>Subject ID | Date of<br>Deviation/<br>Study day | Category | Description |
| xxxxxx/<br>xxxxxx | ddMMMyyyy/<br>xx | Prohibited medication or device | xxxxxxxxxxx |
| | ddMMMyyyy/<br>xx | Assessments and/or procedures/<br>Study treatment supply procedure | xxxxxxxxx |
| xxxxxx/<br>xxxxxxx | ddMMMyyyy/<br>xx | Eligibility criteria not met | xxxxxx |
| xxxxx/<br>xxxxxx | ddMMMyyyy/<br>xx | Not withdrawn after developing withdrawal criteria/<br>Not discontinued from study treatment | xxxxxx |

201893

Protocol: GSK201893
Population: All Treated
Page X of Y

# Listing 7 Listing of Demographic Characteristics

| Center/<br>Subject ID | Year of<br>Birth[1] | Age<br>(Years) | Sex | Child-bearing<br>Potential | Ethnicity | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m^2) |
|---|---|---|---|---|---|---|---|---|
| xxxxx/<br>xxxxxx | xxxx | xx | F | Pre-menarcheal | Hispanic or Latino | xxx.x | xx.x | xx.x |
| xxxxx/<br>xxxxxx | xxxx | xx | F | xxxxxxxxxxx | Not Hispanic or Latino | xxx.x | xx.x | xx.x |
| xxxxx/<br>xxxxxx | xxxx | XX | М | | Not Hispanic or Latino | xxx.x | xx.x | xx.x |

<sup>[1]</sup> For calculating age, birthdate is imputed as June 30 in the year of birth.

# 201893

Protocol: GSK201893
Population: All Treated

Listing 8 Listing of Race

| Center/<br>Subject ID | Race |
|---|---|
| xxxxx/<br>xxxxxx | African American/African Heritage<br>Asian - East Asian Heritage |
| xxxxx/<br>xxxxxx | White - White/Caucasian/European Heritage |
| xxxxx/<br>xxxxxx | African American/African Heritage |

# 201893

Protocol: GSK201893
Population: All Treated

Listing 9 Listing of Family History

| <pre>Treatment = xxxxxx Center/ Subject ID</pre> | A family history of premature coronary artery disease in women <65 yrs or men <55 years in first degree relatives only? |
|---|---|
| / | Voc |
| xxxxx/ | Yes |
| XXXXXX | |
| xxxxx/ | No |
| XXXXXX | |

201893

Protocol: GSK201893
Population: All Treated
Page X of Y

Listing 10 Listing of Medical Conditions

| Treatment = x Center/ | XXXXX | | | NCI CTCAE | |
|---|---|---|---|---|---|
| Subject ID | Category | Medical Condition | Status | Grade | Classification |
| xxxxx/<br>xxxxxx | Cardiovascular<br>Risk Factors | ANGINA PECTORIS | Current | | xxxxx |
| | | DIABETES | Past | | xxxxx |
| | | HYPERTENSION | Current | X | |
| | | | Current | | XXXXX |
| | | | Current | | xxxxxxxxxx |
| | | | Not assessed | | |
| | Other medical condition | xxxxx | Current | | XXXX |
| | | xxxxxx | Past | | xxxx |
| | | xxxxxxxx | Current | X | xxxx |

NCI-CTCAE version 4.03

Programming note: As coding is not done for medical conditions in SDTM MH, please display MHTERM as verbatim term as in other AE listings.

# 201893

Page X of Y Protocol: GSK201893 Population: All Treated

Listing 11 Listing of Disease Characteristics at Initial Diagnosis

| Center/ | Primary<br>Tumor | Date of Diagnosis/ Time Since Diagnosis | Winted and a Common | Histological | Primary<br>Tumor HPV |
|---|---|---|---|---|---|
| Subject ID | Type | (Months) | Histology of Tumor | Grade | Status |
| xxxx/<br>xxxxxx | Bladder | ddMMMyyyy/10.2 | xxxx | Well<br>differentiated | Negative |
| xxxx/ | Xxxx | ddMMMyyyy/xxx.x | XXXX | XXX | XXXXXXX |
| xxxxxx | | | | | |

# 201893

Page X of Y

Protocol: GSK201893 Population: All Treated

Listing 12 Listing of Disease Characteristics at Screening

| Center/<br>Subject ID | Measurable<br>Disease | Non Target<br>Lesions | Stage | Progress on<br>Therapy? | Date of Last<br>Recurrence/Time from<br>Last Recurrence<br>(Months) | Metastatic/<br>Unresectable<br>Disease | Number of<br>Previous<br>Radiotherapy<br>Regimens |
|---|---|---|---|---|---|---|---|
| xxxx/ | Yes | | III | YES | ddMMMyyyy/xx.x | | |
| XXXXXX | | Yes | | | | Yes | 2 |
| xxxx/ | • • | | IIIA | NO | ddMMMyyyy/x.x | | |
| XXXXXX | | • • | | | | XXX | 1 |

201893

Page X of Y Protocol: GSK201893 Population: All Treated

Listing 13

Listing of Prior Anti-Cancer Therapy

Treatment = xxxxxx

| Center/<br>Subject ID | ATC Level 1/<br>Preferred Term/<br>Verbatim Text | Regimen<br>Sequence/<br>Type [1] | Intent | Start Date/<br>Study Day/<br>Stop Date/<br>Study Day | Duration of<br>Therapy<br>(Days) | Small Molecule Targeted<br>Therapy Type |
|---|---|---|---|---|---|---|
| xxxx/<br>xxxxxx | Endocrine & metabolic/<br>Cytoxan/<br>CYTOXAN | 1/<br>C | Neo-Adjuvant | ddMMMyyyy/<br>xxx/<br>ddMMMyyyy/<br>xxx | xxx | AKT Inhibitor |
| | xxxxxxxxx/<br>xxxxxxxxxx/<br>XXXXXXXX | x/<br>H | Induction | ddMMMyyyy/<br>xxx/<br>ddMMMyyyy/<br>xxx | xxx | |

[1] Therapy Type: C=Chemotherapy, H=Hormonal Therapy, I=Immunotherapy, B=Biologic Therapy.

# 201893

Page X of Y

Protocol: GSK201893
Population: All Treated

#### Listing 14 Listing of Prior Anti-Cancer Radiotherapy

| Treatment = xxxxxx | | | | |
|---|---|---|---|---|
| Center/<br>Subject ID | Body Site | Cumulative<br>Dose (unit)/<br>Intent | Start Date/<br>Study Day/<br>Stop Date/<br>Study Day | Duration of<br>Therapy (Days) |
| xxxxxx/<br>xxxxxx | RIGHT UPPER<br>LOBE LUNG | xxx (xxxx)/<br>Local/Regional | ddMMMyyyy/<br>xxx/<br>ddMMMyyyy/<br>xxx | xxx |
| xxxxxx/<br>xxxxxx | CHEST | xxx (xxxx)/<br>Palliative | ddMMMyyyy/<br>xxx/<br>ddMMMyyyy/<br>xxx | xxx |
| xxxxxx/<br>xxxxxx | COLON | xxx (xxxx)/<br>Local/Regional | ddMMMyyyy/<br>xxx/<br>ddMMMyyyy/<br>xxx | xx |
| xxxxxx/<br>xxxxxx | COLON | xxx (xxxx)/<br>Local/Regional | ddMMMyyyy/<br>xxx/<br>ddMMMyyyy/<br>xxx | xx |

# 201893

Protocol: GSK201893 Population: All Treated Page X of Y

Listing 15
Listing of Prior Cancer and Non-Cancer Related Surgical Procedures

| Center | Subject | Classification | Date of<br>Procedure | Study<br>Day | Verbatim Term |
|---|---|---|---|---|---|
| xxxxx | xxxx | Cancer related | ddMMMyyyy | -xx | |
| | | Cancer related | ddMMMyyyy | XX | |
| | xxxx | Cancer related | ddMMMyyyy | XX | |
| xxxxx | xxxx | Cancer related | ddMMMyyyy | -xx | |
| | | Other<br>general | ddMMMyyyy | xxx | Hysterectomy |

201893

Protocol: GSK201893 Population: All Treated Page X of Y

# Listing 16 Listing of Concomitant Medications

| | | Dose/ | | | | |
|---|---|---|---|---|---|---|
| | ATC Level 1/ | Units/ | | | | |
| Center/ | Ingredient/ | Freq/ | Date Started/ | Date Stopped/ | Medication | Reason |
| Subject ID | Verbatim Text | Route | Study Day | Study Day | Category | For Medication |
| xxxxx/ | Fluticasone propionate/ | xx/ | ddMMMyyyy/ | ddMMMyyyy/ | General Concomitant | xxxxx |
| | | | | | Medication | XXXXX |
| XXXXXX | FLIXOTIDE/ | MG/ | XX | XX | Medication | |
| | Asthma | 2XD/ | | | | |
| | | IH | | | | |
| xxxxx/ | XXXXXXXXX/ | xxx/ | ddMMMyyyy/ | ddMMMyyyy/ | Concomitant Medication | XXXXX |
| XXXXXX | XXXXXX | xxx/ | XX | XX | of Interest | |
| | | xxxx/ | | | /Suspected in causing SAE | |
| | | XX | | | | |

201893

Protocol: GSK201893 Population: All Treated Page X of Y

Listing 17

Listing of Blood Products and Blood Supportive Care Products

| Treatment<br>Center/ | = xxxxx<br>For SF, was | | | | | | |
|---|---|---|---|---|---|---|---|
| Subject | it admin- | | | | Quantity o | r | |
| ID | istered? | Product | Product Type | Date | Dose | Unit | Frequency |
| xxxxx/<br>xxxxxx | Р | Blood products | Red Blood Cells | ddMMMyyyy | xxx | | |
| | | | Platelets | ddMMMyyyy | XXX | | |
| | | | Whole Blood | ddMMMyyyy | XXX | | |
| | | | Plasma - FFP | ddMMMyyyy | XXX | | |
| | | | Cryoprecipitate | ddMMMyyyy | XXX | | |
| | | | White Blood Cells | ddMMMyyyy | XXX | | |
| | | | Other Blood Product, specify | ddMMMyyyy | XXX | | |
| | | | | | XXX | | |
| | | Blood supportive care products | darbepoetin alfa (Aranesp) | ddMMMyyyy | XXX | | |
| | | | eltrombopag (i.e. Promacta) | ddMMMyyyy | XXX | | |
| | | | pegfilgrastim (NeulastaR) | ddMMMyyyy | XXX | | |
| | | | romiplostim (i.e. NPlate) | ddMMMvvvv | XXX | | |

SF: stimulating Factor; P = Prophylactically; A = As treatment.

201893

Page X of Y

Protocol: GSK201893

Population: All Treated

# Listing 18 Listing of Follow-Up Anti-Cancer Therapy

Treatment = xxxxxx

| Center/<br>Subject ID | Best Response | Time to<br>Progression<br>(Days) | ATC Level 1/<br>Preferred Term/<br>Verbatim Text | Start Date/<br>Study Day/<br>Stop Date/<br>Study Day | Duration<br>of<br>Therapy | Type<br>of<br>Therapy | Reason for<br>Stopping Therapy |
|---|---|---|---|---|---|---|---|
| xxxx/<br>xxxxxx | Progressive<br>disease | xxx | Endocrine & metabolic/<br>Cytoxan/<br>CYTOXAN | ddMMMyyyy/<br>xxx/<br>ddMMMyyyy/<br>-xxx | xxx d | Chemotherapy | xxxxx |
| | | | xxxxxxxx/<br>xxxxxxxxxxx/<br>xxxxxxxxxxx | ddMMMyyyy/<br>xxx/<br>ddMMMyyyy/<br>-xxx | xxx d | Hormonal | xxxx |
| | | | xxxxxxxx/<br>xxxxxxxxxxx/<br>XXXXXXXXXX | ddMMMyyyy/<br>xxx/<br>ddMMMyyyy/<br>-xxx | xxx d | Radiation | xxxxxxxxxx |

Note: Follow-up surgeries are listed separately.

# 201893

Protocol: GSK201893
Population: All Treated

#### Listing 19 Listing of Follow-Up Surgical Procedures

| Center/<br>Subject ID | Classification | Date of<br>Procedure | Study<br>Day | Verbatim Term |
|---|---|---|---|---|
| xxxxxx/<br>xxxxxx | Cancer related | ddMMMyyyy | xx | |
| | Cancer related | ddMMMyyyy | xx | |
| xxxxxx/ | Cancer related | ddMMMyyyy | xx | |
| xxxxx | Other surgical procedures | ddMMMyyyy | XXX | Hysterectomy |

#### 201893

Protocol: GSK201893 Population: All Treated Page X of Y

Listing 20 Listing of Exposure to GSK2820151

Treatment = xxxxxx

| Center/<br>Subject ID | Average Daily<br>Dose | Start Date/<br>Study Day | Stop Date/<br>Study Day | Dose<br>(mg) | Cumulative<br>Dose<br>(mg) |
|---|---|---|---|---|---|
| xxxx/<br>xxxxxx | xxxx | ddMMMyyyy<br>xx | xx/<br>xx | xx | xx |

Average daily dose is defined as the cumulative dose divided by the duration of exposure for each subject in days. The cumulative dose is the sum of the doses administered for a subject.

Note: Average Daily Dose and Cumulative Dose are derived per subject. Please only display once for each subject.

# 201893

Protocol: GSK201893
Population: All Treated

Listing 21 Listing of Dose Interruptions

| Treatment | _ | XXXXXX |
|-----------|---|--------|

| Center/<br>Subject ID | Dosing Date/<br>Study Day/<br>Dose (mg) | Primary Reason for Interruption/<br>Specify |
|---|---|---|
| xxxxx/<br>xxxxxx | <b>PPD</b> 42/ 0.80 | xxxx/xxxxxxxx |

# 201893

| Protocol: GSK201893 | Page X of Y |
|-------------------------|-------------|
| Population: All Treated | • |

Listing 22 Listing of Dose Reductions

| Center/<br>Subject ID | Dosing Date/<br>Study Day/<br>Dose (mg) | Primary Reason for Reduction/<br>Specify |
|---|---|---|
| xxxxx/<br>xxxxxx | ddMMMyyyy/<br>xx/<br>xx | xxxx/xxxxxxxx |

# 201893

Page X of Y Protocol: GSK201893 Population: All Treated

Listing 23 Listing of Adverse Events Profiles

| Center/<br>Subject<br>ID | Age(Years)/<br>Sex/<br>Race | /<br>Preferred Term/<br>Verbatim Text | Outcome/<br>Onset Date/<br>Resolve Date/<br>Frequency/<br>Duration | Maximum Grade/<br>Serious/<br>Withdrawal from<br>Study | Time since<br>1st Dose/<br>Last Dose | Action(s) taken with Treatment/ Relation to GSK2820151 Treatment | Dose<br>Limiting<br>Toxicity? |
|---|---|---|---|---|---|---|---|
| xxxxx/<br>xxxxxx | 65/<br>Female/<br>White | Nausea/<br>NAUSEA | Resolved/<br>ddMMMyyyy/<br>ddMMMyyyy/<br>Single Episode/<br>xx d | Grade 4/<br>Yes/<br>Yes | xx d/<br>xx d | xxxxxxxxxxxx/<br>XXXX | Yes |

#### 201893

Page X of Y

Protocol: GSK201893 Population: All Treated

Same format for:

Listing 24
Listing of Fatal Serious Adverse Events

Listing 25 Listing of Non-Fatal Serious Adverse Events

Listing 26
Listing of Adverse Events Leading to Discontinuations of GSK2820151 Treatment Profiles

Listing 27
Listing of Adverse Events Leading to Dose Interruptions

Listing 28
Listing of Adverse Events Leading to Dose Reductions

Listing 29
Listing of Adverse Events Recorded as Dose-Limiting Toxicities

Listing 30
Listing of Adverse Events of Special Interest

Programming Note: For Listing 30, Add the following footnote. "Adverse Events of Special Interest are defined as any cardiovascular or death events."

# 201893

Protocol: GSK201893 Population: All Treated Page X of Y

#### Listing 31 Listing of Deaths

| Center/<br>Subject ID | Age(Years)/<br>Sex/<br>Race | Primary Cause of Death/<br>Secondary Cause of Death | Date of Death/<br>Study Day | Time From<br>Last Dose | Last Dose<br>(unit) |
|---|---|---|---|---|---|
| xxxxxx/<br>xxxxxx | 62/<br>M/<br>White | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | ddMMMyyyy/<br>xx | xx d | x/<br>xx |
| xxxxxx/<br>xxxxxx | 45/<br>F/<br>Black | xxxxxxxx/<br>xxxxxxxxxxxx | ddMMMyyyy/<br>xx | xx d | x/<br>xx |
| xxxxxx/<br>xxxxxx | 61/<br>M/<br>South Asian | xxxxxxxx/<br>xxxxxxxxxxxx | ddMMMyyyy/<br>xx | xx d | x/<br>xx |
| xxxxxx/<br>xxxxxx | 52/<br>F/<br>White | xxxxxxxx/<br>xxxxxxxxxxxx | ddMMMyyyy/<br>xx | xx d | x/<br>xx |

# 201893

Protocol: GSK201893 Population: All Treated Page X of Y

#### Listing 32 Listing of Subject Numbers for Specific Causes of Deaths

| Primary Cause of Death | Secondary Cause of Death | Treatment | Number of<br>Subjects | Subject Number |
|---|---|---|---|---|
| Cancer | xxxxxxxxxxxxxxxx | xxxxx<br>xxxxx | 2 | xxxxxx, xxxxxx<br>xxxxxx |
| Myocardial infarction | Haematologic Event | xxxxx | 1 | xxxxxx |

Page X of Y

Protocol: GSK201893
Population: All Treated

Listing 33 Listing of Clinical Chemistry Data

| Center/ | Age(Years)<br>Sex/ | / | Planned | Collection | Study | Converte | ed Data | NR Flag | Grade |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Race | Lab Test (units) | Time | Date | Day | Result | Low-High | [1] | [2] |
| xxxxxx/ | 63/ | Alk Phos (xxx) | Screening | ddMMMyyyy | -x | XX.XX | xx.x- xx.x | | Х |
| XXXXXX | Male/ | | Week 1 Day 1 | ddMMMyyyy | XX | XX.XX | xx.x- xx.x | | X |
| | White | | Week x Day x | ddMMMyyyy | XX | XX.XX | xx.x- xx.x | | X |
| | | | | ddMMMyyyy | XX | XX.XX | xx.x- xx.x | Н | X |
| | | ALT (xxx) | Screening | ddMMMyyyy | -x | XX.XX | xx.x- xx.x | | Х |
| | | | Week 1 Day 1 | ddMMMyyyy | XX | XX.XX | xx.x- xx.x | Н | Х |
| | | | Week x Day x | ddMMMyyyy | XX | XX.XX | xx.x- xx.x | Н | X |
| | | | | ddMMMyyyy | XX | XX.XX | xx.x- xx.x | Н | X |
| | | Hemoglobin (xxx) | Screening | ddMMMyyyy | -x | XX.X | x.x- xx.x | | X |
| | | | Week 1 Day 1 | ddMMMyyyy | XX | XX.X | x.x- xx.x | | X |
| | | | Week x Day x | ddMMMyyyy | XX | XX.X | x.x- xx.x | | X |
| | | | | ddMMMyyyy | XX | XX.X | x.x- xx.x | | X |
| | | Platelets (xxxx) | Screening | ddMMMyyyy | -x | XXX.X | xxx.x-xxx.x | | Х |
| | | | | ddMMMyyyy | XX | XXX.X | xxx.x-xxx.x | | Х |

<sup>[1]</sup> NR for Normal Range flag; H=Above range, L=Below range, N=Normal range.

<sup>[2]</sup> NCI-CTCAE version 4.03

201893

Page X of Y

Protocol: GSK201893 Population: All Treated

Same format for:

Listing 34
Listing of Hematology Data

Listing 35 Listing of Thyroid Function Test Data

> Listing 36 Listing of Urinalysis Data

Listing 37 Listing of Coagulation Data

Listing 38
Listing of Pancreatic Markers Data

Listing 39 Listing of Lipid Panel Data

> Listing 40 Listing of Serum Data

Programming note: for listing 35, please include lab tests as available in SDTM: Thyrotropin (xxx), Thyroxine, Free (pxxx), and Triiodothyronine, Free (xxx).

Programming note for listing 36, please include qualitative urinalysis data (AVALC is populated) per RAP section 11.7. High, Low, NR Flag will be left blank.

201893

Protocol: GSK201893
Population: All Treated
Page X of Y

Listing 41
Listing of Vital Signs

Treatment = xxxxx

| Center/<br>Subject ID | Age(Years)/<br>Sex/<br>Race | Planned<br>Time | Study<br>Day | Actual<br>Date/Time<br>Reading | | Systolic<br>Blood<br>Pressure<br>(mmHg)/<br>Grade | Diastolic Blood Pressure (mmHg)/ Grade | Heart<br>Rate<br>(bests<br>/min) | Respiratory<br>Rate<br>(breaths/min) | Temperature (C) | Weight<br>(kg) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx/<br>xxxxxx | 23/<br>Male/<br>White | Screening<br>Week 1<br>Day 2 | -xx | ddMMMyyyy<br>/hh:mm | 1 | xx/<br>Grade 0 | xx/<br>Grade 0 | хх Н | xx | xx | xx |
| | | | | ddMMMyyyy /hh:mm ddMMMyyyy /hh:mm ddMMMyyyy Average /hh:mm | 3 | xxx/ Grade 1 xxx/ Grade 2 xxx/ Grade 3 | xxx/ Grade 1 xxx/ Grade 2 xxx/ Grade 3 | хх<br>Хх | | | |
| | | Week x Day<br>x | 1 | ddMMMyyyy<br>/hh:mm<br>ddMMMyyyy<br>/hh:mm | | xxx/<br>Grade 3<br>xxx/<br>Grade 0 | xxx/<br>Grade 3<br>xxx/<br>Grade 0 | хх Н | xx<br>xx | хх Н<br>хх Н | xx |
| | | | | ddMMMyyyy<br>/hh:mm | | xxx/<br>Grade 2 | xxx/<br>Grade 2 | xx L | XX | xx L | XX |

Note: L = Low, H = High.

Programming note: repeated readings are only applicable for BP measurements and Heart Rate for some assessments, e.g. Week 1 Day 2.

Systolic BP (mmHg): Grade 0 (<120), Grade 1 (>=120-<140), Grade 2 (>=140-<160) and Grade 3 (>=160), only applies to post-baseline records with increase from baseline.

Diastolic BP (mmHg): Grade 0 (<80), Grade 1 (>=80-<90), Grade 2 (>=90-<100), and Grade 3 (>=100), only applies to post-baseline records with increase from baseline.

Heart Rate (beats/min): L (<60), H (>100), only applies to post-baseline records.

Temperature (C): L (<=35), H (>=38), only applies to post-baseline records.

Protocol: GSK201893
Population: All Treated

Page X of Y

# Listing 42 Listing of ECOG Performance Status Scale

| Center/<br>Subject ID | Age(Years)/<br>Sex/<br>Race | Planned<br>Time | Study<br>Day | Actual<br>Date | ECOG Performance Status * | Change from Baseline |
|---|---|---|---|---|---|---|
| xxx/<br>xxxxxx | 23/<br>Male/<br>White | Screening | -xx | ddMMMyyyy | 1 | |
| | WIIICC | Week x Day x | XX | ddMMMyyyy | 0 | x |
| | | Week x Day x | | | | |

<sup>\*0 =</sup> Fully active, able to carry on all pre-disease performance without restriction;

<sup>1 =</sup> Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work;

<sup>2 =</sup> Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours;

<sup>3 =</sup> Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours;

<sup>4 =</sup> Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair;

<sup>5 =</sup> Dead.

201893

Protocol: GSK201893
Population: All Treated
Page X of Y

Listing 43 Listing of Abnormal ECG Findings

Treatment = xxxxxx
Vendor = ERT

| Center/<br>Subject ID | Age(Years)/<br>Sex/<br>Race | Planned Time/<br>Date/Time/<br>Study Day | Triplicate | Result | Clinically<br>Significant<br>? |
|---|---|---|---|---|---|
| xxx/<br>xxxxxx | 65/<br>White/<br>Female | Week x Day X Pre-dose/<br>ddMMMyyyy<br>hh:mm/ | 1 | Abnormal | No |
| | romaro | x | 2 | Abnormal | No |
| | | | 3 | Abnormal | No |
| xxx/<br>xxxxxx | 58<br>White/<br>Male | Week x Day x 15m/ddMMMyyyy<br>hh:mm/ | X | Abnormal | Yes |

Programming note: ECG labs are collected by both local and central labs. Please display separately.

201893

Protocol: GSK201893
Population: All Treated
Page X of Y

Listing 44 Listing of ECG Values

Treatment = xxxxxx
Vendor = ERT

| Center/<br>Subject ID | Age(Years)/<br>Sex/<br>Race | Planned<br>Time/<br>Date/Time/<br>Study Day | Triplicate | Heart<br>Rate<br>(beats/min.) | PR<br>Interval<br>(msec) | QRS<br>Duration<br>(msec) | QT<br>Interval<br>(msec) | QTc<br>(Fridericia)<br>(msec) |
|---|---|---|---|---|---|---|---|---|
| xxx/<br>xxxxxx | 23/<br>Male/<br>White | Screening Week X Day X Pre-dose | 1<br>2<br>3<br>Average<br>xx | xx<br>xx<br>xx<br>xx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx |

Programming note: ECG labs are collected by both local and central labs. Please display separately.

201893

Protocol: GSK201893 Population: All Treated Page X of Y

Treatment = xxxxxx
Vendor = ERT

| | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|
| Center/<br>Subject ID | Age(Years)/<br>Sex/<br>Race | Planned<br>Time/<br>Date/Time/<br>Study Day | Heart<br>Rate<br>(beats/min.) | PR<br>Interval<br>(msec) | QRS<br>Duration<br>(msec) | QT<br>Interval<br>(msec) | QTc<br>(Fridericia)<br>(msec) |
| xxx/<br>xxxxxx | 23/<br>Male/<br>White | Screening<br>Week X Day X Pre-dose | xx<br>xx | xxx<br>xxx | xxx<br>xxx | xxx | xxx<br>xxx |

Note: Average values of each visit were used to calculate baseline and post-baseline values.

201893

Protocol: GSK201893 Population: All Treated Page X of Y

# Listing 46 Listing of Left Ventricular Ejection Fraction (LVEF) ECHO Results

| Center/<br>Subject ID | Age(Years)/<br>Sex/<br>Race | Planned<br>Time | Study<br>Day | Scan Date | Vendor | LVEF | Absolute Change<br>From Baseline | Scan Results |
|---|---|---|---|---|---|---|---|---|
| xxx/<br>xxxxxx | 23/<br>Male/<br>White | Screening | -x | ddMMMyyyy | VIRTUALSCOPICS | xxx | | Normal |
| | | | | ddMMMyyyy | WAYNE STATE<br>UNIVERSITY<br>PHYSICIAN GROUP | XXX | xxx | Abnormal, Not<br>Clinically<br>Significant |
| | | Week X Day X | | ddMMMyyyy | | XXX | xxx | xxx |

201893

Protocol: GSK201893 Population: All Treated Page X of Y

Listing 47
Listing of Investigator-Assessed Response (RECIST 1.1)

| Center/<br>Subject ID | Measurable<br>Disease at<br>baseline | Planned<br>Time | Date | Resp.<br>Day | Target<br>Lesion<br>Response | Non-Target<br>Lesion<br>Response | New Lesion | Response [1] | If PD, Method of Assessment/ Date [2] |
|---|---|---|---|---|---|---|---|---|---|
| xxxx/<br>xxxxxx | Yes | Screening | ddMMMyyyy | XX | | | | | |
| | | XXXXXXX | ddMMMyyyy | XX | SD | SD | No | SD | |
| | | | ddMMMyyyy | XX | PR | SD | No | PR | |
| | | | ddMMMyyyy | XX | PR | SD | No | PR | |
| | | • • | ddMMMyyyy | XX | PR | SD | No | PD | Radiological |

<sup>[1]</sup> Response: CR = Complete Response, PR = Partial Response, SD = Stable Disease, PD = Progressive Disease, NE = Not Evaluable, NA=Not Applicable.

<sup>[2]</sup> Date provided of non-radiological assessment.

201893

Protocol: GSK201893
Population: All Treated
Page X of Y

Listing 48

Listing of Investigator-Assessed Target Lesions (RECIST 1.1)

Treatment = xxxxxx

| Center/<br>Subject<br>ID | Planned<br>Time | Sum LD (mm)/ Sum Non Lymph Node LD (mm)/ Sum Nadir (mm) | Change in | Percent<br>Change<br>Nadir/<br>Absolute Change<br>Nadir(mm) | Target<br>Lesion<br>Response | Lesion<br>Number | Organ/<br>Location | Method/<br>Slice Thickness/<br>Date/<br>Lesion Assessment Day | LD(mm)[1]/ Target Lesion Status/ Specify the reason |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx/<br>xxxxxx | Screening | xx | | | | 1 | Lung/<br>RIGHT UPPER<br>QUADRANT | CT scan/<br>xx/<br>ddMMMyyyy/<br>xx | xx |
| | | | | | | 2 | Lymph nodes/<br>RIGHT AXILLA | CT scan/<br>xx/<br>ddMMMyyyy/<br>xx | xx |
| | xxxxxxx | xx/<br>xx | xx% | xx%/<br>xx | SD | 1 | Lung/<br>RIGHT UPPER<br>QUADRANT | CT scan/<br>/<br>ddMMMyyyy/<br>xx | xx/<br>Lesion<br>split or<br>divided |
| | | | | | | 2 | Liver/<br>Abdomen | CT scam<br>Xx/<br>ddMMyyy/<br>xx | Xx/<br>Not done/<br>Scan not<br>performed |

<sup>[1]</sup> LD = Lesion diameter

Programming note: Sum of Non Lymph Node LD, Sum of Nadir, and Lesion Status are only collected at post-baseline assessments. For slice thickness, it is only collected at baseline, please retain for post-baseline visits.

# 201893

Protocol: GSK201893 Population: All Treated Page X of Y

Listing 49
Listing of Investigator-Assessed Non-Target Lesions (RECIST 1.1)

| Center/<br>Subject ID | Planned Time | Non-target<br>Lesion<br>Response | Lesion<br>Number | Organ/<br>Location | Method/<br>Date/<br>Lesion Assessment Day | Non-target<br>Lesion Status/<br>Specify the reason |
|---|---|---|---|---|---|---|
| xxxx/<br>xxxxxx | Screening | CR | 1 | Bone/<br>LUMBAR SPINE | MRI/<br>ddMMMyyyy/<br>xx | Present |
| | | | 2 | Bone/<br>THORACIC SPINE | MRI/<br>ddMMMyyyy/<br>xx | Present |
| | | | 3 | Lymph nodes/<br>RIGHT AXILLA | Direct Measure by Physical Exam/ddMMMyyyy/ | Present |
| | Week x Day x | | 1 | Xxx | XX<br>XXX | Not assessable - xxxx |

# 201893

Protocol: GSK201893
Population: All Treated
Page X of Y

# Listing 50 Listing of Investigator -Assessed New Lesions

| Center/ | | | , | Method/ | |
|---|---|---|---|---|---|
| Subject | Planned | Lesion | Organ/ | Date/ | |
| ID | Time | Number | Location | Lesion Assessment Day | Lesion Status |
| PPD | Week 12, | 1 | Lung/ | CT scan/ | Unequivocal |
| | Day 85 | | RIGHT UPPER | PPD | |
| | | | QUADRANT | 172 | |
| | | 2 | Lymph nodes/ | Direct Measure by Physical Exam/ | Unequivocal |
| | | | RIGHT AXILLA | PPD | |
| | | | | 174 | |
| | Week 12, | 1 | Lung/ | CT scan/ | Equivocal |
| | Day 85 | _ | RIGHT UPPER | | nquivocai |
| | Day 05 | | QUADRANT | <b>PPD</b> 181 | |
| | | | QUADRANI | 101 | |
| | Week 24, | 1 | Lung/ | CT scan/ | Unequivocal |
| | Day | | RIGHT UPPER | PPD | |
| | | | OUADRANT | 231 | |

201893

Page X of Y Protocol: GSK201893 Population: All Treated

Listing 51
Listing of Progression Free Survival (RECIST 1.1)

| Center/<br>Subject ID | Age(Years)/<br>Sex/<br>Race | Treatment Start Date/ Event or Censoring Date | Endpoint Description for PFS | PFS (weeks) | New Anti-cancer<br>Therapy Start Date |
|---|---|---|---|---|---|
| xxxxx/ | Female/ | ddMMMyyyy/ | Event: Died | XX.X | ddMMMyyyy |
| XXXXXX | XX | ddMMMyyyy | xx | | 2222 |
| xxxxx/ | Male/ | ddMMMyyyy/ | Censor: xxxxxxxxxxxx | XX.X | |
| XXXXXX | xx | ddMMMyyyy | | | |

201893

Protocol: GSK201893 Page X of Y Population: PK Population

# Listing 52 Listing of GSK2820151 Pharmacokinetic Concentration-Time Data

Treatment = xxxxxx

| Center/<br>Subject ID | Planned<br>Schedule | Planned Time | Date/Actual Time | Time<br>Deviation<br>(Hours) | Actual Relative<br>Time (Hours) | Concentration (ng/mL) |
|---|---|---|---|---|---|---|
| xxx/<br>xxxxxx | Week 1 Day 1 | Pre-dose | ddMMMyyyy/hh:mm | x.xxx | X.XX | NQ |
| | | 15Min post Dose | ddMMMyyyy/hh:mm | | | XXXX.XXX |
| | | 30 Min post Dose | ddMMMyyyy/hh:mm | | | x.xxx |
| | | 1Hour post Dose | ddMMMyyyy/hh:mm | | | xxxx.xxx |
| | | 2Hour post Dose | ddMMMyyyy/hh:mm | | | XXXX.XXX |
| | | 4 Hour post Dose | ddMMMyyyy/hh:mm | | | xxxx.xxx |

NQ = Non-quantifiable.

201893

Protocol: GSK201893 Page X of Y Population: PK Population

Listing 53
Listing of Derived GSK2820151 Pharmacokinetic Parameters

| Center/ | Cmax | tmax | AUC(0-t) | AUC(0-tau) | AUC(0-inf) | t1/2 | C tau | Ro [1] | CL/F | Vz/F |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | (ng/mL) | (h) | (h*ng/mL) | (unit) | (h*ng/mL) | (h) | (unit) | | (mL/h) | (mL) |
| xxx/<br>xxxxxx | xx.xx | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |

<sup>[1]</sup> Ratio of AUC(0-tau): AUC(0-tau) on Week 3 Day 4/AUC(0-tau) on Week 1 Day 1